CLINICAL TRIAL: NCT06336135
Title: A Prospective, Single-blind, Randomized, Placebo-controlled, Clinical Trial Evaluating Reduction in Severity and Duration of Symptoms After Laser Therapy With Acorn aHFS
Brief Title: Reduction in Symptoms After Laser Therapy With Acorn aHFS
Status: Completed | Type: Observational
Sponsor: Acorn Biolabs Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-001
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Skin Aging
Keywords: skin, aging, rejuvenation, laser resurfacing, autologous secretome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: autologous hair follicle derived secretome — aHFS is a cosmetic topical intended to be applied to the human body after skin resurfacing cosmetic procedures. aHFS is produced from the plucked hair follicles of each individual, making it autologous.
  Other Names: Acorn autologous hair follicle secretome; aHFS

SUMMARY:
This study evaluates the severity and duration of symptoms experienced after laser therapy comparing four post-procedure topical products. Each product is applied to an individual region of interest (5 cm diameter) on the back or décolleté according to randomization code after laser therapy. The subject, blind to the product applied to each of 4 regions of interest, assesses eight symptoms daily for 14 days. Photography is performed daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age: ≥18 and ≤60 years
* Any skin tone Fitzpatrick score 1-2 (light), 3-4 (medium), 5-6 (dark)
* Competent and willing to provide written, informed consent to participate in all study activities

Exclusion Criteria:

* Pregnant women
* Are participating/have participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by Sponsor
* Use of retinoids 7 days prior to the procedure
* Active cutaneous infections in the treatment area
* Diseases that could inhibit healing, such as scleroderma, or other cutaneous conditions that could confound study results
* Subjects unable to communicate with the investigator and staff
* Any health condition that in the investigator's opinion should preclude participation in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are healthy adults receiving laser skin rejuvenation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Reduction in severity and duration of symptoms | 2 weeks
  Each region of interest will be evaluated daily for the severity and duration of eight symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Campbell, PhD, Study Director — Acorn Biolabs Inc.
Locations (1):
- Rejuuv Medi Spa, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.